CLINICAL TRIAL: NCT05322473
Title: Phase 2, Randomized, Parallel-group, Double-blind, Placebo-controlled Study of Sonelokimab in Patients With Active Moderate to Severe Hidradenitis Suppurativa
Brief Title: Evaluation of Sonelokimab for the Treatment of Patients With Active Moderate to Severe Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1095-HS-201
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration; Adalimumab; Anti-Inflammatory Agents; Sonelokimab; Nanobody; Folliculitis; Apocrine Gland Disease; Acne Inversa
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration; Folliculitis | interventions — sonelokimab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- sonelokimab dose 1 (Experimental): Subjects randomized to this arm will receive assigned sonelokimab dosage regimen and placebo to maintain the blinding with adalimumab and placebo arms during the Treatment Period.
  Interventions: Drug: Sonelokimab (M1095)
- sonelokimab dose 2 (Experimental): Subjects randomized to this arm will receive assigned sonelokimab dosage regimen and placebo to maintain the blinding with adalimumab and placebo arms during the Treatment Period.
  Interventions: Drug: Sonelokimab (M1095)
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo during the Double-Blind Treatment Period and will be re-randomized to receive a sonelokimab dosage regimen during Part B.
  Interventions: Other: Placebo
- adalimumab (Active Comparator): Subjects randomized to this arm will receive adalimumab during the Double-Blind Treatment Period and will be reallocated to receive sonelokimab dosage regimen during Part B.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Sonelokimab (M1095) — randomized treatment; parallel-group
  Arms: sonelokimab dose 1; sonelokimab dose 2
Drug: Adalimumab — randomized treatment; parallel-group
  Arms: adalimumab
Other: Placebo — randomized treatment; parallel-group
  Arms: Placebo

SUMMARY:
This is a study to demonstrate the clinical efficacy and safety of the nanobody® sonelokimab administered subcutaneously (sc) compared with placebo in the treatment of adult participants with moderate to severe hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥18 years of age;
2. Participant has been diagnosed with hidradenitis suppurativa as determined by the investigator and has a history of signs and symptoms of hidradenitis suppurativa dating back at least 6 months prior to the Screening Visit;
3. Participant has a total abscess and/or inflammatory nodule (AN) count of ≥5;
4. Participant has hidradenitis suppurativa lesions present in ≥2 distinct anatomical areas, at least one of which must contain single or multiple fistulas (i.e., be Hurley Stage II or III);
5. Participant had an inadequate response to appropriate systemic antibiotics for treatment of hidradenitis suppurativa (or demonstrated intolerance to, or had a contraindication to, systemic antibiotics for treatment of their HS), in the investigator's opinion;
6. Participant must be, in the opinion of the investigator, at both the Screening Visit and study treatment initiation, a suitable candidate for treatment with adalimumab per approved local product information.

Exclusion Criteria:

1. Participants with known hypersensitivity to sonelokimab or any of its excipients;
2. Participants with known hypersensitivity to adalimumab or any of its excipients;
3. Participant has a draining fistula count of ≥20 at the Screening Visit;
4. Participant has any other active skin disease or condition that may, in the opinion of the investigator, interfere with the assessment of hidradenitis suppurativa;
5. Prior exposure to more than 2 biologic response modifiers;
6. Participant has a diagnosis of ulcerative colitis or Crohn's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response 75 | Week 12
  Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 75 (HiSCR75), where HiSCR75 is defined as at least a 75% reduction from baseline in abscess and inflammatory nodule (AN) count, with no increase from baseline in abscess or draining fistula count.

SECONDARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response 50 | Week 12
  Proportion of participants achieving HiSCR50
Change in International Hidradenitis Suppurativa Severity Score System | Week 12
  Change from baseline in International Hidradenitis Suppurativa Severity Score System (IHS4)
  The IHS4 score is calculated as follows: number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild, 4 to 10 signifies moderate and 11 or higher signifies severe disease.
Dermatology Life Quality Index (DLQI) | Week 12
  Proportion of participants achieving a Dermatology Life Quality Index (DLQI) total score of ≤5
  The DLQI produces a numeric score that can range from 0 to 30. A higher score indicates greater health-related quality of life impairment.
Reduction from Numerical Rating Scale (NRS30) in Patient's Global Assessment of Skin Pain (PGA Skin Pain) | Week 12
  Proportion of participants achieving at least 30% reduction and at least 2-unit reduction from Baseline in Numerical Rating Scale (NRS30) in Patient's Global Assessment of Skin Pain (PGA Skin Pain) among subjects with Baseline NRS ≥3
  The NRS is a numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Kristian Reich, M.D., Ph.D. (equ.), Study Director — MoonLake Immunotherapeutics AG
Locations (51):
- United States (15):
  - Clinical Site, Fountain Valley, California
  - Clinical Site, Los Angeles, California
  - Clinical Site, Miami, Florida
  - Clinical Site, Ormond Beach, Florida
  - Clinical Site, St. Petersburg, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Beverly, Massachusetts
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Omaha, Nebraska
  - Clinical Site, New York, New York
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Charleston, South Carolina
  - Clinical Site, Nashville, Tennessee
  - Clinical Site, Bellaire, Texas
- Bulgaria (2):
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
- Canada (10):
  - Clinical Site, Calgary, Alberta
  - Clinical Site, Winnipeg, Manitoba
  - Clinical Site, Fredericton, New Brunswick
  - Clinical Site, St. John's, Newfoundland and Labrador
  - Clinical Site, Hamilton, Ontario
  - Clinical Site, London, Ontario
  - Clinical Site, Markham, Ontario
  - Clinical Site, Newmarket, Ontario
  - Clinical Site, Peterborough, Ontario
  - Clinical Site, Saskatoon, Saskatchewan
- Germany (12):
  - Clinical Site, Bad Bentheim
  - Clinical Site, Berlin
  - Clinical Site, Bochum
  - Clinical Site, Darmstadt
  - Clinical Site, Dresden
  - Clinical Site, Frankfurt
  - Clinical Site, Hamburg
  - Clinical Site, Kiel
  - Clinical Site, Lübeck
  - Clinical Site, Mahlow
  - Clinical Site, München
  - Clinical Site, Münster
- Clinical Site, Dublin, Ireland
- Netherlands (2):
  - Clinical Site, Bergen op Zoom
  - Clinical Site, Rotterdam
- Poland (9):
  - Clinical Site, Gdansk
  - Clinical Site, Krakow
  - Clinical Site, Lodz
  - Clinical Site, Olsztyn
  - Clinical Site, Ossy
  - Clinical Site, Ostrowiec Świętokrzyski
  - Clinical Site, Poznan
  - Clinical Site, Warsaw
  - Clinical Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No